CLINICAL TRIAL: NCT07027917
Title: The Impact of Virtual Reality Application on Pain, Anxiety, and Vital Parameters During Pleural Catheter Insertion: A Randomized Controlled Trial
Brief Title: The Application of Virtual Reality Goggles During Pleural Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Almira Gurcan, Uzman hemşire, Adnan Menderes Üniversitesi, Cerrahi Hastalıkları Hemşireliği Anabilim Dalı, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-97594401-804.01-455320
Record Dates: First submitted 2025-02-20; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pain; Catheter (Other)
Keywords: pain; anxiety; nursing; pleural catheter; virtual reality; vital signs; state anxiety; VAS; VR
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Goggles During Catheterization (Experimental): In this group, virtual reality glasses were applied during the pleural catheter insertion procedure.
  Interventions: Device: Virtual Reality Goggles
- Standard Catheterization Without VR (No Intervention): No additional intervention was applied to this group other than the routine catheter insertion procedure.

INTERVENTIONS:
Device: Virtual Reality Goggles — VR
  Arms: Virtual Reality Goggles During Catheterization

SUMMARY:
The aim of this study is to examine the effects of virtual reality glasses applied to individuals who will undergo pleural catheter placement on pain, anxiety, and vital parameters. The main research questions that the study aims to answer are as follows:

* Does the application of virtual reality goggles have an effect on pain measured during pleural catheter insertion?
* Does the application of virtual reality goggles have an effect on anxiety measured during pleural catheter insertion?
* Does the application of virtual reality goggles have an effect on the vital parameters measured during pleural catheter insertion?

The researcher compared the intervention and control groups to determine whether the glasses have an effect on the measurable parameters (pain, anxiety, and vital signs).

DETAILED DESCRIPTION:
Today, both pharmacological and non-pharmacological methods are used to reduce patients' pain and anxiety during invasive procedures. Distraction techniques hold an important place among non-pharmacological methods. Virtual reality (VR) glasses can be effective in reducing perceived pain and anxiety by allowing patients to divert their attention elsewhere during procedures.

This study was conducted to evaluate the distribution of virtual reality brightness on patients' pain and anxiety levels.

The study was designed as a randomized controlled trial by the researchers. The patients included in the study were divided into two groups: the intervention group (exposed to virtual reality) and the control group (standard care). Following stratified randomization, randomization was carried out using a simple random number table.

Application:

During the insertion phase, Shinecon brand virtual reality glasses were placed on the patients during the connection process, and underwater images were shown.

During routine phases, no distraction method was applied, and only the procedure was followed.

All patients' vital signs (blood pressure, heart rate, oxygen saturation) were recorded before, during, and after the procedure. Pain levels were assessed using the Visual Analog Scale (VAS) before and after the procedure. Additionally, anxiety levels were measured using the State-Trait Anxiety Inventory (STAI-S, STAI-T) before and after the procedure.

This study supports the use of virtual reality technology as a non-pharmacological intervention to improve patient comfort during minimally invasive procedures and provides evidence-based information.

ELIGIBILITY:
Inclusion Criteria:

Written or verbal consent to participate, Being over 18 years of age, Not having any psychiatric diagnosis, Not having any problems with vision, hearing, perception or communication.

Exclusion Criteria:

Being unconscious Experiencing pain due to any other problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Pain severity | From immediately before to 10 minutes after catheter insertion
  Pain severity will be assessed using the Visual Analog Scale (VAS), a 10 cm scale ranging from 0 (no pain) to 10 (worst possible pain), measurements will be taken before, during and after pleural catheter insertion.

SECONDARY OUTCOMES:
Anxiety level | From immediately before to 10 minutes after catheter insertion
  Anxiety will be measured using the State-Trait Anxiety Inventory (STAI). The inventory consist of 20 items rated on a 4 point Likert scale ranging from 1 (not at all), to 4 (very much so). The state anxiety subscale will be pre and post intervention to evaluate changes in situational anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes Üniversitesi, Aydin, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes